CLINICAL TRIAL: NCT06838988
Title: Ultrasonographic Patterns and Pathological Correlation in the Diagnosis of Subcutaneous Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suthinee Rutnin, Suthinee Rutnin, MD, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MURA2025/83
Record Dates: First submitted 2025-02-11; First posted 2025-02-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Nodules; Ultrasonography; Panniculitis
Keywords: Nodules; Ultrasonography; panniculitis
MeSH Terms: conditions — Panniculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Transcutaneous ultrasonography (Experimental): This is a single group study with one intervention arm where every subjects received ultrasonographic evaluations of their skin lesions (subcutaneous nodules)
  Interventions: Diagnostic Test: Transcutaneous ultrasound

INTERVENTIONS:
Diagnostic Test: Transcutaneous ultrasound — The ultrasonographic characteristics of the subcutaneous nodules were evaluated using an ultrasound machine (Venue Go™, wide-band linear array ultrasound probe (hockey stick shape), frequency range between 6.7 MHz and 18.0 MHz, from GE HealthCare Illinois, United States).
  The procedure for capturing images at the location of the lesion of interest is as follows:
  * Brightness mode (B-mode): Record at least 4 images using a depth of 2 cm.
  * Color Doppler mode: Record images along the vertical axis (1 image) and along the horizontal axis (1 image). The two axes mentioned above must be perpendicular to each other.
  * Video recording: Capture at least 10 seconds of video in both Brightness mode and Color Doppler mode.

SUMMARY:
The objective of this study is to explore the role of ultrasonography (non-invasive imaging device) in the diagnosis of subcutaneous nodules (mass/bumb underneath the skin).

Patients who presented with subcutaneous nodules and was indicated for diagnostic skin biopsies were recruited. Prior to skin biopsies (not part of the study's intervention), ultrasonography(intervention) was used to examine the characteristics of the nodules. The ultrasonographic findings are then compared to the pathological results to explore the role of ultrasonography in differentiating each disease or group of diseases that presented with skin nodules.

DETAILED DESCRIPTION:
Panniculitis refers to a group of conditions involving inflammation of the fat cells in the subcutaneous tissue. It can result from various causes, such as inflammation, infection, vasculitis (inflammation of blood vessels), or lymphoproliferative disorders (abnormal lymphocyte proliferation). In general, it is challenging to determine the cause of subcutaneous tissue inflammation based solely on skin manifestations, as patients often present with similar symptoms, such as subcutaneous lumps, tenderness, and redness, usually found in the lower limbs. Therefore, diagnosis often requires a comprehensive patient history taking, physical examinations, and sometimes biopsy for histopathological examination to confirm the diagnosis. Occasionally, additional tests, including immunohistochemistry, cultures, or polymerase chain reaction (PCR), may be necessary for greater diagnostic accuracy.

Since 1997, Ackerman has proposed diagnostic guidelines for panniculitis based on histopathological findings, initially categorizing it according to the site of inflammation into septal panniculitis and lobular panniculitis. Further classification considers whether vasculitis is present. However, even with physical examination and histopathological analysis, accurately classifying panniculitis remains challenging. In 2007, Requena and colleagues highlighted limitations in biopsy, such as the selection of lesions with differing characteristics or lesions at different stages, resulting in varying histopathological features. Moreover, the depth or insufficient amount of tissue collected for biopsy may reduce diagnostic accuracy.

Since 1979, medical advancements have led to the increased use of ultrasound in dermatological diagnosis. Low-frequency ultrasound machines (2 MHz) were initially used to examine skin lesions, such as skin inflammation or subcutaneous nodules. In 1983, Miyauchi and colleagues began using higher-frequency ultrasound (10 MHz) to study ultrasound characteristics compared to histopathological results in patients presenting with subcutaneous or dermal nodules. Over time, the use of higher-frequency ultrasound became more common, as it provides better detail and convenience, being a simple, safe, and cost-effective procedure.

For panniculitis, research has shown that ultrasound can assist in diagnosis. In 2020, Romani and colleagues studied the correlation between ultrasound findings and histopathology in 62 cases of panniculitis. Septal panniculitis typically shows thickening of the septa with hypoechoic areas resembling a jigsaw pattern, difficult to compress, increased blood flow, and possible clotting in veins. Lobular panniculitis shows hyperechoic fat with irregular borders, without septal thickening or increased vascularity, and may show fat necrosis or extension into muscles and adjacent tissues. However, further research is needed for clear differentiation between types of panniculitis based on ultrasound features.

Subsequent studies have used ultrasound to describe various forms of panniculitis, including those caused by gout, erythema nodosum, lupus erythematosus, and subcutaneous T-cell lymphoma, among others.

In conclusion, diagnosing panniculitis in patients with subcutaneous nodules remains challenging and relies on a combination of physical examination, patient history, histopathology, and sometimes additional tests like immunohistochemistry, cultures, or PCR. These diagnostic procedures can lead to unnecessary testing and delays in diagnosis. Ultrasound data can assist in selecting appropriate laboratory tests, facilitate diagnosis and treatment monitoring, and aid in selecting biopsy sites. However, there is no comprehensive collection of ultrasound data for different conditions, which is why this study was conducted to gather this information and explore the correlation between ultrasound findings and histopathological features for more accurate diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older who presented with subcutaneous nodules
* Indicated for pathological examination for disease diagnosis.
* Patients with subcutaneous nodules located in areas where a tissue sample can be taken down to the fat layer.
* Patients who agree to participate in the project by signing the consent form.

Exclusion Criteria:

* Presence of inflammation or other tumors that can mimic panniculitis, such as painful lipomas, cellulitis, and leg interstitial edema.
* Patients with diseases that significantly alter the structure of the skin or subcutaneous tissue, such as scleroderma or severe edema.
* A history of previous treatments in the area of the subcutaneous mass (e.g., surgery, radiation therapy, or high-dose steroid treatment) that may interfere with ultrasound results.
* Patients with lesions on the head or mucous membranes of the body.
* Pregnant or breastfeeding patients.
* Presence of wounds or open sores in the area to be examined with ultrasound.
* A history of coagulopathy (blood clotting disorders).
* Patients with metal implants in the area of interest that may interfere with ultrasound imaging.
* Participants who refuse or withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Subcutaneous echogenicity | Through study completion averaging 2 years
  In this study, we aim to explore the relationship between ultrasonographic characteristics of subcutaneous nodules(A) and the pathological findings from biopsy samples(B).
  (A) The primary outcome measure is the subcutaneous echogenicity A1) hyper-echoic, A2) hypo-echoic, A3) iso-echoic.
  (B) Pathological results are graded as either B1) Infectious, B2) Non-infectious

SECONDARY OUTCOMES:
Subcutaneous fat septum thickness | Through study completion averaging 2 years
  In this study, we aim to explore the relationship between ultrasonographic characteristics of subcutaneous nodules (A) and the pathological findings from biopsy samples (B).
  (A) The secondary outcome measure is the subcutaneous fat septum thickness A1) more than or equal to 1mm : septal thickening present, A2) less than 1mm : septal thickening absent
  (B) Pathological results are graded as either B1) Infectious, B2) Non-infectious

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospital, Bangkok, Ratchathewi, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang BS, Choi SH, Cha HJ, Jung YK, Lee JH, Jeong AK, Shin SH, Kwon WJ. Subcutaneous panniculitis-like T-cell lymphoma: US and CT findings in three patients. Skeletal Radiol. 2007 Jun;36 Suppl 1:S67-71. doi: 10.1007/s00256-006-0173-6. Epub 2006 Aug 15. PMID 16909278
- [Background] Nazzaro G, Maronese CA, Passoni E. Ultrasonographic diagnosis of erythema nodosum. Skin Res Technol. 2022 Mar;28(2):361-364. doi: 10.1111/srt.13112. Epub 2021 Nov 23. No abstract available. PMID 34813122
- [Background] Delgado-Jimenez Y, Fraga J, Garcia-Diez A. Infective panniculitis. Dermatol Clin. 2008 Oct;26(4):471-80, vi. doi: 10.1016/j.det.2008.05.005. PMID 18793979
- [Background] Gaviria JL, Ortega VG, Gaona J, Motta A, Medina Barragan OJ. Unusual Dermatological Manifestations of Gout: Review of Literature and a Case Report. Plast Reconstr Surg Glob Open. 2015 Aug 10;3(7):e445. doi: 10.1097/GOX.0000000000000420. eCollection 2015 Jul. PMID 26301134
- [Background] Maldonado Cid P, Rubio Flores C, Prats Caelles I, Leis Dosil VM, Alfageme Roldan F, Richi Alberti P, Santonja Garriga C, Diaz Diaz RM. High-frequency ultrasound features in a case of gouty panniculitis. Dermatol Online J. 2017 Jun 15;23(6):13030/qt33j2z14m. PMID 28633741
- [Background] Romani J, Giavedoni P, Roe E, Vidal D, Luelmo J, Wortsman X. Inter- and Intra-rater Agreement of Dermatologic Ultrasound for the Diagnosis of Lobular and Septal Panniculitis. J Ultrasound Med. 2020 Jan;39(1):107-112. doi: 10.1002/jum.15080. Epub 2019 Jun 27. PMID 31245860
- [Background] Catalano O, Wortsman X. Dermatology Ultrasound. Imaging Technique, Tips and Tricks, High-Resolution Anatomy. Ultrasound Q. 2020 Dec;36(4):321-327. doi: 10.1097/RUQ.0000000000000520. PMID 33298770
- [Background] Wortsman X, Alfageme F, Roustan G, Arias-Santiago S, Martorell A, Catalano O, Scotto di Santolo M, Zarchi K, Bouer M, Gonzalez C, Bard R, Mandava A, Gaitini D. Guidelines for Performing Dermatologic Ultrasound Examinations by the DERMUS Group. J Ultrasound Med. 2016 Mar;35(3):577-80. doi: 10.7863/ultra.15.06046. Epub 2016 Feb 17. PMID 26887446
- [Background] Nessi R, Betti R, Bencini PL, Crosti C, Blanc M, Uslenghi C. Ultrasonography of nodular and infiltrative lesions of the skin and subcutaneous tissues. J Clin Ultrasound. 1990 Feb;18(2):103-9. doi: 10.1002/jcu.1870180207. PMID 2156901
- [Background] Mandava A, Ravuri PR, Konathan R. High-resolution ultrasound imaging of cutaneous lesions. Indian J Radiol Imaging. 2013 Jul;23(3):269-77. doi: 10.4103/0971-3026.120272. PMID 24347861
- [Background] Gropper CA, Stiller MJ, Shupack JL, Driller J, Rorke M, Lizzi F. Diagnostic high-resolution ultrasound in dermatology. Int J Dermatol. 1993 Apr;32(4):243-50. doi: 10.1111/j.1365-4362.1993.tb04261.x. No abstract available. PMID 8486453
- [Background] Requena L. Normal subcutaneous fat, necrosis of adipocytes and classification of the panniculitides. Semin Cutan Med Surg. 2007 Jun;26(2):66-70. doi: 10.1016/j.sder.2007.02.001. PMID 17544956
- [Background] Requena L, Sanchez Yus E. Panniculitis. Part II. Mostly lobular panniculitis. J Am Acad Dermatol. 2001 Sep;45(3):325-61; quiz 362-4. doi: 10.1067/mjd.2001.114735. PMID 11511831
- [Background] Requena L, Yus ES. Panniculitis. Part I. Mostly septal panniculitis. J Am Acad Dermatol. 2001 Aug;45(2):163-83; quiz 184-6. doi: 10.1067/mjd.2001.114736. PMID 11464178